CLINICAL TRIAL: NCT05826665
Title: Observational Study to Examine the Procedural and Outcomes of AF Ablation Assisted by STAR Apollo™ Mapping System
Status: Recruiting | Type: Observational
Sponsor: Kansas City Heart Rhythm Research Foundation (Other)
Collaborators: Kansas City Heart Rhythm Institute (Other); St. Bernards Medical Center (Unknown); Sarasota Medical Center (Unknown)
Responsible Party: Sponsor
Other Study IDs: KCHRRF_Star Apollo_0018
Record Dates: First submitted 2023-04-12; First posted 2023-04-24 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- STAR Apollo Mapping System Group: Patients who have been referred for persistent AF catheter ablation, who have already had AF recurrence post Pulmonary Vein Isolation (PVI), will be considered for this study.
  Interventions: Other: Persistent AF ablation assisted with the STAR Apollo Mapping System

INTERVENTIONS:
Other: Persistent AF ablation assisted with the STAR Apollo Mapping System — This exploratory hypothesis generating data set will be collected during standard AF ablation procedures using FDA cleared technologies as described in their Instructions for Use (IFU). No randomization or experimental protocols will be used during this study, and all follow up will be performed as per the center's standard of care(SOC).

SUMMARY:
STAR Apollo Mapping System is an FDA cleared mapping technology that can analyze the signals collected during the ablation procedure on the 3D mapping system and give the physician further insight into the AF activation patterns which may assist them in identifying areas responsible for maintaining Atrial Fibrillation (AF). The STAR Apollo Mapping System system allows clinicians, after treating the Pulmonary Veins (PV), to collect data from the atria during clinical AF procedures using standard FDA cleared catheters and devices. This study aims to examine the impact of the STAR Apollo Mapping System on procedural and acute outcomes in a multicenter observational study.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common heart rhythm abnormality. It affects 1 in 100 people. It can cause unpleasant symptoms of palpitation, shortness of breath and in some can cause heart failure or stroke. AF is triggered by abnormal electrical signals originating both in the pulmonary veins (PV), the veins that drain blood from the lungs into the heart, and in the rest of the left atrium, the heart chamber that the PVs drain into. AF can be successfully treated by a procedure called catheter ablation. This involves passing a wire up the vein at the top of the leg and delivering radiofrequency energy to the atrial tissue. This renders that tissue electrically inert. For many years this procedure has been guided by 3D cardiac mapping systems capable of showing the position of the catheters in the heart and recording their electrical signals. By doing a series of radiofrequency treatments around the mouth of the PVs it is possible to electrically isolate them so that PV signals cannot start or sustain AF. This leaves the left atrial signals untreated and limits the success of the procedure to 50%. To date clinicians have tried numerous ways to identify these remaining left atrial signals, but so far, their efforts have not improved the outcomes of ablation over just isolating the PVs alone (50% success rate). STAR Apollo Mapping System is an FDA cleared mapping technology that can analyze the signals collected during the ablation procedure on the 3D mapping system and give the physician further insight into the AF activation patterns which may assist them in identifying areas responsible for maintaining AF. The STAR Apollo Mapping System system allows clinicians, after treating the PVs, to collect data from the atria during clinical AF procedures using standard FDA cleared catheters and devices. This study aims to examine the impact of the STAR Apollo Mapping System on procedural and acute outcomes in a multicenter observational study.

ELIGIBILITY:
Inclusion Criteria:

* Indication for ablation of persistent AF
* Age >18 years
* Persistent AF >7 days and total continuous duration <2 years
* Patients have previously undergone pulmonary vein isolation, using any technique and have had AF recurrence.
* Patients have limited additional ablation at their first procedure (e.g. right atrial flutter line).

Exclusion Criteria:

* Patients with previous ablation in more than one region of the left atrium in addition to the pulmonary veins.
* Patients with longstanding persistent AF (continuous duration >2 years) or significant substrate (mitral valve disease, scarring, very dilated atria >50mm).
* Creatinine clearance estimated glomerular filtration rate (eGFR) <30mls/min
* Contraindication to anticoagulation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been referred for persistent AF catheter ablation, who have already had AF recurrence post PVI, will be considered for this study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-10-02 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
To determine the impact of STAR Apollo Mapping System on the procedural parameters of persistent AF ablation | 12 Months
  The primary objective for the study is to determine the impact of STAR Apollo Mapping System on the procedural parameters of persistent AF ablation. These include procedure duration and the number of radiofrequency (RF) lesions applied post PVI.

SECONDARY OUTCOMES:
To observe the acute procedural outcomes and the features of the STAR Apollo Mapping System data | 12 Months
  The secondary objective is to observe the acute procedural outcomes and the features of the STAR Apollo Mapping System data and the physician's treatment plan that may influence outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Dhanunjaya Lakkireddy, MD, Principal Investigator — Kansas City Heart Rhythm Institute
Locations (4):
- United States (4):
  - St.Bernards Medical Center, Jonesboro, Arkansas
  - Sarasota Medical Center, Sarasota, Florida
  - Kansas City Heart Rhythm Institute - Roe Clinic, Overland Park, Kansas
  - Overland Park Regional Medical Center, Overland Park, Kansas